CLINICAL TRIAL: NCT04193371
Title: Department of Traditional Chinese Medicine (TCM), Peking University Third Hospital, Beijing, China
Brief Title: Effects of Acupuncture on Body Mass Index in Overweight and Obese Women With Polycystic Ovary Syndrome (PCOS )
Acronym: PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PekingUTH TCM
Record Dates: First submitted 2019-11-06; First posted 2019-12-10 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-03

CONDITIONS: PCOS; Overweight; Obesity
Keywords: PCOS; Overweight; Obesity; Acupuncture; Lifestyle management
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional case-control part and an open-labelled RCT with a comparative effectiveness design. The inter-ventions to be tested are (1) acupuncture during 4 months+lifestylemanagement; (3) sham acupuncture+lifestyle management
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active acupuncture + lifestyle management (Experimental): Participants in this group are treated by active acupuncture and lifestyle management for 4 months and follow up 4 months after the last treatment.
  Interventions: Other: Active acupuncture; Other: Lifestyle management
- control acupuncture + lifestyle management (Sham Comparator): Participants in this group are treated by control acupuncture and lifestyle management for four months and follow up 4 months after the last treatment.
  Interventions: Other: Sham acupuncture; Other: Lifestyle management

INTERVENTIONS:
Other: Active acupuncture — The rationale of the active acupuncture protocol is based on Western Medical Acupuncture theories and follows CONSORT and STRICTA protocols. All patients received acupuncture treatment for 30 minutes three times a week, with a maximum of 48 acupuncture treatments.
  Arms: active acupuncture + lifestyle management
Other: Sham acupuncture — In the sham acupuncture protocol, 2 needles were inserted superficially to a depth of less than 5 mm, 1 in each shoulder and 1 in each upper arm at nonacupuncture and non-meridian points, and then, 4 needles were attached to electrodes and the stimulator was turned on to mimic the active acupuncture but with zero intensity, no electrical stimulation. They also received the treatment for 30 minutes three times a week and a maximum of 48 treatments.
  Arms: control acupuncture + lifestyle management
Other: Lifestyle management — All women will receive lifestyle management before randomization after baseline measurements. The lifestyle management assisted by a PCOS lifestyle management system (Invention patent, ZL 2015 1 0500978.9).
  All participants will get a step-counter for daily use and physical exercise diary for daily reporting of exercise: number of steps, type of activity, intensity and time (minutes). Once a week each participant receive a SMS in which they report the activity during the week.

SUMMARY:
This is a cross-sectional case-control study combined with a randomised controlled trial (RCT) study. This study aims to compare the effect of acupuncture, with usual care (lifestyle management) for weight control, with BMI (Body Mass index) as main outcome along with improvement of reproductive and metabolic dysfunction in overweight and obese women with PCOS, and further exploring the alteration of lipidomics, bile acid omics, proteomics and branched-chain amino acids between PCOS and the normal controls, and before and after the acupuncture treatment in different gourps.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) affects 6 to 18% of all women and is the most common female endocrine and metabolic disorder during the reproductive years. PCOS is characterized by anovulation, hyperandrogenism and metabolic dysfunction.Obesity is ~40% higher in women with PCOS than in healthy women. Overweight results in irregular cycles, insulin resistance and infertility. Acupuncture is assumed to reduce weight The overall hypothesis is that if the Body mass index (BMI) decreased, ovulation can be induced, hyperandrogenism decreased, and insulin sensitivity improved in these women. Although several treatment strategies have shown efficacy, importantly, there is a need for Comparative Effectiveness Research (CER) to strengthen the evidence base for clinical and policy decision-making. Therefore, the investigators aim to compare the effect of acupuncture, with usual care (lifestyle management) for weight loss, and improvement and prevention of reproductive and metabolic dysfunction in overweight and obese women with PCOS. We further compare the differences of PCOS and the controls with the methods of lipidomics, bile acid omics, proteomics and branched-chain amino acids, exploring the mechanisms of acupuncture on PCOS with this kind of methods.

ELIGIBILITY:
Inclusion Criteria: PCOS

* Age 20 to 40 years
* BMI≥ 24 to <40
* PCOS diagnosis according to Rotterdam criteria 2003 with at least two of the following three symptoms: (1) infrequent ovulation or anovulation; (2) hyperandrogenism or clinical manifestations of high blood androgen; (3) ultrasound findings of polycystic ovaries in 1 or 2 ovaries, or ≥12 follicles measuring 2 to 9 mm in diameter, and/or ovarian volume ≥10 mL.

Inclusion criteria: Controls

Controls should have BMI>25to<40, regular cycles with 28 days±2 days and no signs of hyperandrogenism and PCO morphology on ultrasound

Exclusion Criteria:

* Exclusion of other endocrine disorders such as androgen secreting tumors, suspected Cushing's syndrome and non-classic congenital adrenal hyperplasia (17-hydroxyprogesterone < 3nmol/L) thyroid dysfunction and hyperprolactinemia.
* Type I diabetes or not well controlled type II diabetes
* Pharmacological treatment (cortizone, antidepressant, other antidiabetic treatment such as insulin and acarbose, hormonal contraceptives, hormonal ovulation induction or other drugs judged by discretion of investigator) within 12 weeks. Depo Provera or similar within 6 months.
* Pregnancy or breastfeeding the last 6 months
* Acupuncture last 3 months
* Daily smoking and alcoholic intake

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — No, the enrollment is based on biological sex
Enrollment: 106 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | After 4 months of intervention;
  PCOS's weight in kilograms divided by the square of her height in meters, reported in kg/m2

SECONDARY OUTCOMES:
total body fat | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with a body composition analyzer (Tanita Corporation, model MC-180, Japan) .
body fat and lean ratio | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with a body composition analyzer (Tanita Corporation, model MC-180, Japan) .
visceral fat | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with a body composition analyzer (Tanita Corporation, model MC-180, Japan) .
basal metabolic rate | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with a body composition analyzer (Tanita Corporation, model MC-180, Japan) .
antral follicle count | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined the ovarian morphology with the B-ultrasound
sex hormone binding globulin (SHBG) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
anti-mullerian hormone (AMH) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
follicle stimulating hormone (FSH) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
luteinizing hormone (LH) | After 4 months of intervention Follow-up 4 months after last treatment.，
  examined with the blood sample
Progestin (P) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Estrogen (E2) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Androgen(T) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Androstenedione (A2) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
HOMA-IR | After 4 months of intervention， Follow-up 4 months after last treatment.
  will be assessed during the oral glucose tolerance test (OGTT) , calculation of HOMA-IR: [fasting insulin (μU/mL) × fasting glucose (mmol/L)] / 22.5)
HOMA- β | After 4 months of intervention， Follow-up 4 months after last treatment.
  will be assessed during the oral glucose tolerance test (OGTT) ,calculation of HOMA-β: 20 × fasting insulin (mU/mL) / (fasting plasma glucose (mmol/L) - 3.5
glycated hemoglobin ( HbA1c) | After 4 months of intervention， Follow-up 4 months after last treatment.
  The insulin and glucose response in blood
total cholesterol | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
triglycerides | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
high density lipoprotein (HDL) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
low density lipoprotein (LDL) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
lipometabonomic/lipidomics | After 4 months of intervention， Follow-up 4 months after last treatment.
  Detection with the method of metabonomic in blood, the sample size is about 20 participants in each group.
bile acid omics | After 4 months of intervention， Follow-up 4 months after last treatment.
  Detection with the method of metabonomic in blood, the sample size is about 20 participants in each group
β-endorphin | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
5- hydroxytryptamine (5-HT) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
FerrimanGallwey (FG )value | After 4 months of intervention， Follow-up 4 months after last treatment.
  To determine changes in women's hairy with FG rating scale (0-36 score), the higher, the worse.
short form-36 (SF36) | After 4 months of intervention， Follow-up 4 months after last treatment.
  determine the health quality of life by the questionnaire of SF36 (0-100 score), the higher, the better.
EuroQol health index scale (EQ-5D) | After 4 months of intervention， Follow-up 4 months after last treatment.
  determine the health quality of life by the questionnaire of EQ-5D (0-100 score), the higher, the better.
polycystic ovary syndrome questionnaire (PCOSQ); | After 4 months of intervention， Follow-up 4 months after last treatment.
  determine the Effects of PCOS specific symptoms on the participants by the questionnaire of and polycystic ovary syndrome questionnaire (PCOSQ)(26-182 score); the higher, the better.
Self-Rating Anxiety Scale (SAS) | After 4 months of intervention， Follow-up 4 months after last treatment.
  determine the anxiety level with the questionnaire of SAS (20-100 score), the higher, the worse.
Self-Rating Depress Scale (SDS) | After 4 months of intervention， Follow-up 4 months after last treatment.
  determine the depress level with the questionnaire of SDS (20-100 score), the higher, the worse.
Body mass index (BMI) | Follow-up 4 months after last treatment.
  Weight in kilograms divided by the square of her height in meters, reported in kg/m2
Fibroblast growth factor 19(FGF-19) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Ghrelin | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Interleukin 6( IL-6 ) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Interleukin 8( IL-8 ) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Interleukin 22( IL-22 ) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Tumor Necrosis Factor-Alpha (TNF-α) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Gamma-Amino Butyric Acid(GABA) | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
dopamine（DA） | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
Glutamate | After 4 months of intervention， Follow-up 4 months after last treatment.
  examined with the blood sample
proteomics | After 4 months of intervention
  Detection with the Proteomic techniques in blood, the sample size is about 30 participants in each group.
branched-chain amino acids | After 4 months of intervention
  examined with the blood sample, the sample size is about 30 participants in each group.

CONTACTS AND LOCATIONS:
Overall Officials: haolin zhang, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes